## **Title Page**

#### **Protocol Title:**

A Phase 2, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of BNC210 Compared to Placebo for the Acute Treatment of Social Anxiety Disorder

**Protocol Number: BNC210.013** 

**Amendment Number: 1** 

Compound: BNC210

**Brief Title:** A Phase 2 Study of BNC210 for the Acute Treatment of Social Anxiety Disorder

**Study Phase: 2** 

**Sponsor Name:** Bionomics Limited

Legal Registered Address: 200 Greenhill Road, Eastwood, SA, 5063, AUSTRALIA

**Regulatory Agency Identifier Number(s):** 

Registry ID
IND
NCT

**Approval Date: 17-NOV-2021** 

#### **Confidentiality Statement**

This document contains the confidential information of **Bionomics Limited**. It is provided to you as an Investigator or consultant for review by you, your personnel, and the applicable Institutional Review Board (IRB). Your acceptance of this document constitutes an agreement that you will not disclose the information contained herein to others without the prior written consent of **Bionomics Limited**, unless it is necessary to obtain informed consent from potential study participants. No other use or reproduction is authorized by **Bionomics Limited**, nor does **Bionomics Limited** assume any responsibility for unauthorized use of this protocol.

Sponsor Signatory:



**Bionomics Limited** 

## **Protocol Amendment Summary of Changes Table**

| DOCUMENT HISTORY | | |
|---|---|---|
| Document | Date | Rationale for Amendment |
| Original Protocol<br>Version 1.0 | 30-Sep-2021 | Not applicable |
| Protocol Version 1.1 | 17-Nov-2021 | |

## **Table of Contents**

| 7 |
|----------|
| 7 |
| 11 |
| 13 |
| 14 |
| 14 |
| 15 |
| 15 |
| 17 |
| 18 |
| 21 |
| 21 |
| 21 |
| 23 |
| 24 |
| 24 |
| 25 |
| 27 |
| 27 |
| 20 |
| 28 |
| 29 |
| 29 |
| 30 |
| 31 |
| 32<br>32 |
| 32 |
| 32 |
| 33 |
| 33 |
| 35 |
| 35 |
| 35 |

| 7.3. | Lost to Follow-up. | 35 |
|---|---|---|
| 8. | Study Assessments and Procedures | 36 |
| 8.1. | Efficacy Assessments | 37 |
| 0.1.2 | | 2.7 |
| 8.1.2. | Subjective Units of Distress Scale (SUDS) | |
| 8.1.3. | Spielberger State-Trait Anxiety Inventory (STAI) | |
| 8.1.4. | Self-Statements During Public Speaking (SSPS) | |
| 8.2. | Safety Assessments | |
| 8.2.1. | Physical Examinations | |
| 8.2.2. | Vital Signs | |
| 8.2.3. | Electrocardiograms | |
| 8.2.4.<br>8.2.5. | Clinical Safety Laboratory Assessments | |
| | Suicidal Ideation and Behavior Risk Monitoring | 39 |
| 8.3. | Adverse Events (AEs), Serious Adverse Events (SAEs), and | 40 |
| 8.3.1. | Other Safety Reporting Time Period and Frequency for Collecting AE and SAE | 40 |
| 0.3.1. | | 40 |
| 8.3.2. | Information | |
| 8.3.3. | - The state of the | |
| 8.3.4. | Follow-up of AEs and SAEs. | |
| 8.3.5. | Regulatory Reporting Requirements for SAEs | |
| 8.4. | Plasma Bioanalysis | |
| 8.5. | Genetics | |
| 8.6. | Biomarkers | |
| 8.7. | Immunogenicity Assessments. | |
| 8.8. | Medical Resource Utilization and Health Economics | |
| 0.0. | | |
| 9. | Statistical Considerations | |
| 9.1. | Statistical Efficacy Hypotheses | |
| 9.1.1. | Multiplicity Adjustment | |
| 9.2. | Analysis Sets | |
| 9.3. | Statistical Analyses | |
| 9.3.1. | | 44 |
| 9.3.2. | Study Participants and Demographics | |
| 9.3.3. | Primary Endpoint(s)/Estimand(s) Analysis | |
| 9.3.4. | Secondary and Exploratory Endpoints Analysis | 46 |
| 9.4. | Interim Analysis | 16 |
| J.T. | mornii / mary 515 | <del>4</del> 0 |
| 10. | Supporting Documentation and Operational Considerations | 47 |
| 10.1. | Appendix 1: Regulatory, Ethical, and Study Oversight | ••••• <del>•</del> / |
| 10.1. | Considerations | 17 |
| 10.1.1. | Regulatory and Ethical Considerations | |
| 10.1.1. | Financial Disclosure | |
| 10.1.2. | Informed Consent Process | |
| 10.1.3. | Data Protection. | 48 |

| 10.1.5. | Data Quality Assurance | 49 |
|---------|-----------------------------------------------------------|----|
| 10.1.6. | Source Documents | |
| 10.1.7. | Study and Site Closure | 50 |
| 10.1.8. | Publication Policy | 50 |
| 10.2. | Appendix 2: Clinical Laboratory Tests | 51 |
| 10.3. | Appendix 3: AEs and SAEs: Definitions and Procedures for | |
| | Recording, Evaluating, Follow-up, and Reporting | 53 |
| 10.3.1. | Definition of AE | |
| 10.3.2. | Definition of SAE | 54 |
| 10.3.3. | Recording and Follow-Up of AE and/or SAE | 55 |
| 10.3.4. | Reporting of SAEs | 58 |
| 10.4. | Appendix 4: Contraceptive and Barrier Guidance | |
| 10.4.1. | Definitions | 60 |
| 10.4.2. | Contraception Guidance | 61 |
| 10.5. | Appendix 5: Liver Safety: Suggested Actions and Follow-up | |
| | Assessments | 62 |
| 10.6. | Appendix 6: Abbreviations | 64 |
| 11. | References | 67 |

#### 1. Protocol Summary

#### 1.1. Synopsis

Protocol Title: A Phase 2, Randomized, Double-blind Study to Evaluate the Efficacy and

Safety of BNC210 Compared to Placebo for the Acute Treatment of Social

**Anxiety Disorder** 

**Brief Title:** A Phase 2 Study of BNC210 for the Acute Treatment of Social Anxiety

Disorder

#### **Rationale:**

This Phase 2 study will assess the potential efficacy of BNC210 in the acute treatment of social anxiety disorder (SAD). Anxiety symptoms in adults with SAD will be evaluated during an induced public speaking challenge following single-dose acute administration of BNC210 (or placebo).

Previous human studies with BNC210 have established its safety and tolerability and demonstrated statistically significant results in a Phase 1 study using a panic model in healthy volunteers and in a Phase 2a study in patients with generalized anxiety disorder (GAD).

| _ |
|---|

Objectives and Endpoints, and Estimands:

| Objectives | Endpoints |
|---|---|
| Primary | |
| To assess the effects of BNC210 compared to placebo in reducing self-reported anxiety severity as measured by the Subjective Units of Distress Scale (SUDS) in the performance phase of a public speaking challenge | The difference in change in SUDS scores after oral administration of a single dose of BNC210 or placebo from baseline to the average of the performance phase of a public speaking challenge |
| Secondary | |
| To assess the effects of BNC210 compared to placebo in reducing self-reported anxiety severity as measured by the SUDS in a public speaking challenge | The difference in change in SUDS scores after oral administration of a single dose of BNC210 or placebo from baseline to the performance phase of a public speaking challenge |
| To assess the effects of BNC210 compared to placebo in reducing self-reported symptoms of anxiety as measured by the Spielberger State-Trait Anxiety Inventory - State component (STAI-State) in a public speaking challenge | <ul> <li>The difference in change in SUDS scores after oral administration of a single dose of BNC210 or placebo from baseline to the anticipation phase of a public speaking challenge</li> <li>The difference in change in STAI-</li> </ul> |
| To assess the effects of BNC210 compared to placebo in reducing self-reported negative cognitions during speaking as measured by the Self- | State scores after oral administration of a single dose of BNC210 or placebo from baseline to the performance phase of a public speaking challenge |
| Statements During Public Speaking Scale (Negative Self-Statements subscale; SSPS-N) in a public speaking challenge To assess the safety and tolerability of | <ul> <li>The difference in change in STAI-<br/>State scores after oral administration<br/>of a single dose of BNC210 or<br/>placebo from baseline to the<br/>anticipation phase of a public</li> </ul> |
| BNC210 | <ul> <li>The difference in change in SSPS-N scores after oral administration of a single dose of BNC210 or placebo from baseline to the performance phase of a public speaking challenge</li> </ul> |
| | <ul> <li>The difference in change in SPSS-N<br/>scores after oral administration of a<br/>single dose of BNC210 or placebo</li> </ul> |



#### Overall Design:

This is a randomized, double-blind, placebo-controlled, 3-arm, parallel-group, multi-center study comparing the effects of single acute doses of BNC210 and placebo when participants with SAD perform an induced public speaking challenge. Participants will attend a Screening Visit to confirm eligibility. Approximately 150 participants who fulfill the inclusion criteria and none of the exclusion criteria will return to the clinic within 14 days after the Screening Visit and be randomized to receive either 225 mg BNC210, 675 mg BNC210, or matched placebo (in a ratio of 1:1:1). Randomized participants will then receive a single oral dose of their allocated study intervention and approximately 1 hour later, will each participate in a public speaking challenge. Approximately 1 week post speaking challenge, a follow-up assessment will be conducted by phone/video conference for any reports of AEs.

#### **Brief Summary:**

The purpose of this study is to assess the effects of an acute dose of BNC210 compared to p lacebo on reducing the severity of anxiety levels provoked by a public speaking challenge and measured using the SUDS in patients with SAD.

#### **Number of Participants:**

Approximately 250 participants will be screened to achieve a total enrollment of approximately 150 randomly assigned participants.

#### **Intervention Groups and Duration:**

The total duration for each participant enrolled in the study is expected to be approximately 3 weeks following the sequence below:

- Screening Period: 14 days (+3)
- Treatment Period with public speaking challenge: 1 day
- Follow-up Period:  $7 (\pm 3)$  days after treatment

Details of study assessments to be conducted at each visit are included in the Schedule of Activities (SoA) in Sections 1.3 and 1.4.

Each participant will be randomized in a 1:1:1 ratio to receive a single dose of 225 mg BNC210, 675 mg BNC210, or placebo. Treatment assignments will be double-blinded.



## 1.3. Schedule of Activities (SoA) - Overview

| | | | Treat | ment Day | | Follow-up |
|---|---|---|---|---|---|---|
| ASSESSMENTS <sup>1</sup> | Screening ≤ 14 days (+3 days) | Baseline / Pre-Dose <sup>2</sup> | Dosing | Public<br>Speaking<br>Challenge | Post-<br>Challenge | via phone/video<br>conference<br>7 days post<br>treatment<br>(±3 days) |
| Informed consent | X | | | | | , , , |
| Inclusion and exclusion criteria <sup>3</sup> | X | X | | | | |
| Demography | X | | | | | |
| Medical history including current & prior medications | X | | | | | |
| Structured Clinical Interview for DSM-5 Disorders - Clinical Trials version (SCID-5-CT) | X | | | | | |
| Liebowitz Social Anxiety Scale (LSAS) | X | | | | | |
| Hamilton Depression Rating Scale (HAM-D) | X | | | | | |
| Columbia-Suicide Severity Rating Scale (C-SSRS) <sup>4</sup> | X | X | | | | |
| Human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg) and Hepatitis C virus (HCV) antibody screen | X | | | | | |
| Serum pregnancy test (if applicable) | X | | | | | |
| Urine drug screen <sup>5</sup> | X | X | | | | |
| Physical examination <sup>6</sup> | X | X | | | | |
| Vital signs <sup>7</sup> | X | X | | | X8 | |



| | | | Trea | tment Day | | Follow-up |
|---|---|---|---|---|---|---|
| | Screening ≤ 14 days | Baseline / | | Public<br>Speaking | Post- | via phone/video conference 7 days post treatment |
| ASSESSMENTS <sup>1</sup> | (+3 days) | Pre-Dose <sup>2</sup> | Dosing | Challenge | Challenge | (±3 days) |
| 12-lead electrocardiogram (ECG) <sup>9</sup> | X | | | | X <sup>10</sup> | |
| Clinical laboratory tests (hematology, biochemistry, urinalysis) | X | X | | | X <sup>11</sup> | |
| Concomitant medications recording | X | X | | | | |
| Urine pregnancy test (if applicable) <sup>12</sup> | | X | | | | |
| Randomization <sup>13</sup> | | X | | | | |
| Subjective Units of Distress Scale (SUDS) <sup>14</sup> | | X | | X | X | |
| Spielberger State-Trait Anxiety Inventory-State component (STAI-State) <sup>15</sup> | | X | | X | X | |
| Self-Statements During Public Speaking () (SSPS) <sup>16</sup> | | X | | X | X | |
| Dosing with Study Intervention <sup>17</sup> | | | X | | | |
| Blood sample collection for BNC210 concentration <sup>18</sup> | | | | | X | |
| Assessment of participant's readiness for discharge <sup>19</sup> | | | | | X | |
| Adverse Event (AE) recording | | | X | $X^{20}$ | X | X |



## 1.4. Schedule of Activities (SoA) - Efficacy Assessments on Treatment Day

| | | | | | Public Speaking Challenge | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline / Pre-Dose | | Pre-Dose Restin | Resting / Post-Dose | | Speech Preparation - Anticipation Phase (2 mins duration) | | Performance Phase<br>(5 mins duration) | | | | | |
| | prior to<br>dosing) | Dosing | (~55 mins post dose) | on<br>Challenge | 0<br>min | 1<br>min | 2<br>min | 0<br>min | 1<br>min | 2<br>min | 3<br>min | 4<br>min | 5<br>min |
| Subjective Units of<br>Distress Scale (SUDS) | X | | X | | X | x | X | X | X | x | X | X | X |
| Spielberger State-Trait<br>Anxiety Inventory –<br>State component<br>(STAI-State) | X | | X | | | | x | | | | | | х |
| Self-Statements<br>During Public<br>Speaking (SSPS) <sup>1</sup> | X | | X | | | | х | | | | | | х |

#### 2. Introduction

Bionomics Limited is developing BNC210 for the treatment of anxiety disorders and traumaand stressor-related disorders. BNC210 is a negative allosteric modulator of the alpha-7 nicotinic acetylcholine receptor (alpha-7 nAChR), which represents a novel target for the treatment of these disorders. BNC210 is a new chemical entity that has exhibited potent anxiolytic activity in a range of animal models at low doses with a wide therapeutic window. There is an absence of adverse effects, particularly those associated with treatments for acute anxiety disorders, such as benzodiazepines, and the antidepressants used in first-line pharmacotherapy for chronic anxiety disorders.

#### 2.1. Study Rationale

This Phase 2 study will assess the potential benefits of BNC210 in the acute treatment of social anxiety disorder (SAD). Anxiety symptoms in adults with SAD will be evaluated during a public speaking challenge, following single-dose acute administration of 1 of 2 dosages of BNC210 or placebo.

Previous human studies with BNC210 have established its safety and tolerability and demonstrated statistically significant results in a Phase 1 study using a panic model in healthy volunteers and in a Phase 2a study in patients with generalized anxiety disorder (GAD).

| _ |
|---|

## 2.2. Background

#### 2.2.1. Disease Background

Social Anxiety Disorder is a serious anxiety disorder characterized by the persistent, intense fear of social or performance-related situations in which an individual is exposed to unfamiliar people or to possible scrutiny by others. Social Anxiety Disorder can also manifest from specific triggers such as a fear of public speaking or be induced by social interactions across any variety of situations. Those suffering from SAD often fear that they will act in a way or show anxiety symptoms that will be embarrassing and humiliating, thus further inducing anxiety. This fear can affect work, school, and other day-to-day activities and can even make it hard to develop and maintain friendships. Most cases of SAD develop in adolescence or early adulthood and without treatment can persist and prevent individuals from reaching their full potential.

Antidepressants, including selective serotonin reuptake inhibitors (SSRIs) and serotonin noradrenaline reuptake inhibitors (SNRIs), currently serve as first-line pharmacotherapies for SAD. However, SSRIs/SNRIs typically require several weeks of chronic administration before onset of action, making them inadequate for the treatment of acute anxiety episodes in SAD. There are no approved drugs for the acute treatment of SAD, although anti-anxiety medications such as benzodiazepines, or beta blockers which help reduce the physical symptoms of anxiety, are commonly used off-label. Benzodiazepines are potent, fast-acting anxiolytic drugs, but they are sedating and carry significant safety risks, including memory and motor impairment, serious risk of abuse, addiction, physical dependence, and withdrawal reactions, as highlighted in the FDA Drug Safety Communication, September 2020. Those with SAD are also at increased risk of alcohol use disorder, turning to alcohol and other substances in anticipation of social situations.

Thus, there is a need for improved therapeutics for acute treatment of SAD, with fast onset of action and fewer side effects, which might be achieved by targeting a different mechanism of action.

| <br> |
|------|

| i |
|---|
| 1 |
| _ |
| _ |
| ı |
| _ |
| _ |



## 2.3. Benefit/Risk Assessment

More detailed information about the known and expected benefits and risks and reasonably expected AEs of BNC210 can be found in the Investigator's Brochure (IB) and the participant Informed Consent Form (ICF).

No potential significant risks have been identified in the nonclinical or clinical studies of BNC210. At this stage in development, the benefit-risk profile of BNC210 appears favorable.

## 3. Objectives, Endpoints, and Estimands

| Objectives | Endpoints |
|---|---|
| Primary | |
| To assess the effects of BNC210 compared to placebo in reducing self-reported anxiety severity as measured by the Subjective Units of Distress Scale (SUDS) in the performance phase of a public speaking challenge | The difference in change in SUDS scores after oral administration of a single dose of BNC210 or placebo from baseline to the average of the performance phase of a public speaking challenge |
| Secondary | |
| To assess the effects of BNC210 compared to placebo in reducing self-reported anxiety severity as measured by the SUDS in a public speaking challenge | The difference in change in SUDS scores after oral administration of a single dose of BNC210 or placebo from baseline to the performance phase of a public speaking challenge |
| <ul> <li>To assess the effects of BNC210 compared to placebo in reducing self-reported symptoms of anxiety as measured by the Spielberger State-Trait Anxiety Inventory - State component (STAI-State) in a public speaking challenge</li> <li>To assess the effects of BNC210 compared to placebo in reducing self-reported negative cognitions during speaking as measured by the Self-Statements During Public Speaking Scale (Negative Self-Statements subscale; SSPS-N) in a public speaking challenge</li> <li>To assess the safety and tolerability of BNC210</li> </ul> | <ul> <li>The difference in change in SUDS scores after oral administration of a single dose of BNC210 or placebo from baseline to the anticipation phase of a public speaking challenge</li> <li>The difference in change in STAI-State scores after oral administration of a single dose of BNC210 or placebo from baseline to the performance phase of a public speaking challenge</li> <li>The difference in change in STAI-State scores after oral administration of a single dose of BNC210 or placebo from baseline to the anticipation phase of a public speaking challenge</li> <li>The difference in change in SSPS-N scores after oral administration of a single dose of BNC210 or placebo from baseline to the performance phase of a public speaking challenge</li> </ul> |
| | <ul> <li>The difference in change in SPSS-N<br/>scores after oral administration of a<br/>single dose of BNC210 or placebo<br/>from baseline to the anticipation phase<br/>of a public speaking challenge</li> </ul> |



## **Primary Estimand**

The primary efficacy endpoint of mean change in the SUDS score from baseline to the average across all timepoints in the performance phase of a public speaking challenge will be compared between the placebo and the BNC210 groups.



## 4. Study Design

## 4.1. Overall Design

This is a randomized, double-blind, placebo-controlled, 3-arm, parallel-group, multi-center study c omparing the effects of single acute doses of BNC210 and placebo when participants with SAD perform an induced public speaking challenge. Participants will attend a Screening Visit to confirm eligibility. Approximately 150 participants who fulfill the inclusion criteria and none of the exclusion criteria will return to the clinic within 14 days after the Screening Visit and be randomized to receive either 225 mg BNC210, 675 mg BNC210, or matched placebo (in a ratio of 1:1:1). Randomized participants will then receive a single dose of their allocated study intervention and approximately 1 hour later, each will participate in a public speaking challenge. Approximately 1 week later, a follow-up assessment will be conducted by phone/video conference for any reports of AEs.

Protocol BNC210.013

Details are included in the Schedule of Activities (SoA), Section 1.3 and 1.4).

## 4.2. Scientific Rationale for Study Design

The primary objective of this study is to assess the effects of BNC210 compared to placebo on public speaking anxiety symptom severity using the SUDS, a commonly used scale for measuring performance anxiety in behavioral avoidance tasks such as a public speaking challenge. A public speaking challenge is a very consistent experimental model for the induction of anxiety in both healthy volunteers and in individuals diagnosed with SAD or social phobia, and has been used in studies investigating the effects of pharmacological and nonpharmacological interventions on subjective measures of anxiety in patients with SAD

A double-blind, placebo-controlled study design has been chosen as a well-established and appropriate study design to minimize the potential for bias in study assessments or in reporting of AEs. Clinic staff and participants are blinded to treatment assignments to ensure objective reporting. In addition, participants will be randomized 1:1:1 to receive 1 of 2 doses of BNC210 or placebo to ensure there are no order effects and to further minimize bias.





## 4.4. End of Study Definition

The end of the study is defined as the date of the follow-up assessment for the last participant in the study.

#### 5. Study Population

Investigators will be responsible for evaluating potential participants against the study eligibility criteria during the Screening Period. At the initial Screening Visit, each participant will participate in the informed consent process and sign and date the ICF before any procedures specified in this protocol are performed.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

#### 5.1. Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

#### Age

1. Participant is 18 to 65 years of age (inclusive) at the time of signing informed consent.

#### **Type of Participant and Disease Characteristics**

- 2. Participant has a current diagnosis of SAD as defined in the Diagnostic and Statistical M anual of Mental Disorders, fifth edition (DSM-5) and confirmed by the Structured Clinical Interview for DSM-5 Disorders Clinical Trials version (SCID-5-CT).
- 3. Participant has a Liebowitz Social Anxiety Scale (LSAS) total score of ≥70 and a subscore of 3 on Question 6 (Fear or Anxiety subscale) at Screening.
- 4. In the opinion of the Investigator, the participant has a high probability for adherence with and completion of the study.
- 5. Participant is fluent in English and able to understand and comply with written and verbal protocol-related requirements.
- 6. Participant is able to swallow tablets.

#### **Sex and Contraceptive/Barrier Requirements**

- 7. Participants' contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
  - a. Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 60 days after the dose of study intervention:
    - Refrain from donating sperm PLUS, either:
      - Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent

OR

 Must agree to use a male condom with female partner using an additional highly effective contraceptive method with a failure rate of < 1% per year as described in Appendix 4: Contraceptive and Barrier Guidance, when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant

- b. Female participants are eligible to participate if they are not pregnant or breastfeeding and the following conditions apply:
  - Is of nonchildbearing potential (WONCBP) as defined in Appendix 4:
     Contraceptive and Barrier Guidance.

OR

- o Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of < 1% per year), preferably with low user dependency, as described in Appendix 4: Contraceptive and Barrier Guidance during the study intervention period and for at least 60 days after the dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The Investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of study intervention.
- A WOCBP must have a negative serum pregnancy test at Screening and a negative urine test at baseline (within 24 hours before the first dose of study intervention).

The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

#### **Informed Consent**

8. Capable of giving signed informed consent as described in Appendix 1: Regulatory, Ethical, and Study Oversight Considerations which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

#### 5.2. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

#### **Medical Conditions**

- 1. Participant has a history of schizophrenia, bipolar disorder, or psychotic disorders as identified at Screening, or has a current <u>clinically predominant</u> diagnosis of any other Axis I disorder, other than SAD, at the time of the Screening Visit.
- 2. Participant has a score of ≥18 on the Hamilton Rating Scale for Depression (HAM-D) at Screening.
- 3. Participant has moderate or severe alcohol-use disorder, or any other substance-use disorder (any severity), according to DSM-5, in the 12 months prior to Screening.
- 4. Participant has increased risk of suicide, defined as:
  - Any suicide attempt in the 12 months prior to Screening disclosed by the participant using the Columbia-Suicide Severity Rating Scale (C-SSRS).

- Any suicidal ideation with intent (yes to item 4 and/or 5) or suicidal behavior in the past 12 months, as captured at Screening using the C-SSRS.
- 5. Participant has presence of impaired renal function as indicated by clinically significant abnormal creatinine, blood urea nitrogen (BUN), or plasma urea, or moderate to severe renal dysfunction as defined by the Cockcroft-Gault equation (estimated glomerular filtration rate [eGFR] <50 mL/min).
- 6. Participant has alanine transaminase (ALT), aspartate transaminase (AST) or alkaline phosphatase (ALP) >2.0 × upper limit of normal (ULN).
- 7. Participant has total bilirubin  $>1.5 \times ULN$  (isolated bilirubin  $>1.5 \times ULN$  is acceptable if total bilirubin is fractionated and direct bilirubin <35%).
- 8. Participant has current or chronic history of liver disease. This includes, but is not limited to, hepatitis virus infections, drug- or alcohol-related liver disease, nonalcoholic steatohepatitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, α-1 antitrypsin deficiency, primary biliary cholangitis, primary sclerosing cholangitis, or any other liver disease considered clinically significant by the Investigator.
- 9. Participant has any clinically significant abnormalities in laboratory test results (biochemistry, hematology, or urinalysis) as assessed by the Investigator.
- 10. Participant has blood pressure systolic >160 mmHg or diastolic >90 mmHg. Two repeat measures are allowed at the discretion of the Investigator.
- 11. Fridericia-corrected QT interval (QTcF) >450 msec for males and QTcF >470 msec for females, or QTc >480 msec in participants with bundle branch block, as measured by ECG at Screening.
- 12. Participant has any clinically significant ECG abnormality as determined by the Investigator at Screening.
- 13. Participant has a family history of congenital long QT syndrome, Brugada syndrome, or unexplained sudden cardiac death.

#### **Prior/Concomitant Therapy**

- 14. Participant has used psychotropic medications, including antidepressants, mood stabilizers, stimulants, antipsychotics, anticonvulsant drugs (including gabapentinoids), hypnotics (zolpidem, zopiclone, eszopiclone, zaleplon), acetylcholinesterase inhibitors, or anxiolytics such as benzodiazepines within 30 days of Screening. Participants who have been taking benzodiazepines daily within 90 days of Screening are also not eligible to participate. No concurrent use of these medications is allowed on study.
- 15. Participant has used beta blockers, doxazosin, prazosin, clonidine, first-generation sedating H1 antihistamines, any recreational drugs, over-the-counter medication, or herbal preparations to treat symptoms of anxiety or SAD within 30 days of Screening. No concurrent use of these medications is allowed on study.
- 16. Participant has used cytochrome P450 3A4 inducers within 30 days of Screening.
- 17. Participant has used moderate-strong cytochrome P450 3A4 inhibitors within 2 weeks of Screening. This includes, but is not limited to, grapefruit or grapefruit-containing products.

#### **Prior/Concurrent Clinical Study Experience**

- 18. Participant is currently enrolled OR has previously participated in another investigational study in which an investigational intervention (e.g., drug, vaccine, invasive device) was administered within 30 days before signing of consent in this clinical study.
- 19. Participant has previously participated in a study that involved a public speaking challenge.

#### **Diagnostic Assessments**

- 20. Participant has a positive result for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) at Screening.
- 21. Participant has a positive urine test for an illicit substance, including cannabis. No concurrent use of these substances is allowed on study.

#### Other Exclusions

- 22. Participant has a history of allergies, allergic reactions, or hypersensitivity to BNC210 or its excipients.
- 23. Participants who, in the opinion of the Investigator, are not suitable to participate in the study due to clinically significant findings from medical history that could interfere with the objectives of the study or put the participant at risk or any other reason the Investigator deems applicable.

## **5.3.** Lifestyle Considerations

There are no specific lifestyle considerations or restrictions applicable to this study outside of the criteria detailed in Sections 5.1, 5.2, and 6.8.

#### 5.4. Screen Failures

Participants who sign and date the ICF but who fail to meet the inclusion and exclusion criteria are considered screen failures. Reason(s) for screen failure must be documented by the Investigator and provided to the Sponsor in a timely fashion.

A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any SAEs.

In the event that a participant fails a clinical laboratory or ECG screening assessment, that assessment can be repeated once only during the Screening Period. The repeat assessment must be completed within the allowed Screening Period (14 days) for eligibility purposes. If the repeat assessment cannot be completed within the Screening Period, the participant must be re-screened in entirety. Participants who fail any other screening assessment must be screen-failed.

Individuals who do not meet the criteria for participation in this study (screen failure) may be rescreened, if deemed appropriate by the Investigator and with prior approval from the sponsor/medical monitor. Rescreened participants should be reconsented and be assigned a new participant number (Subject ID) for every screening/rescreening event.

# 5.5. Criteria for Temporarily Delaying Randomization or Administration of Study Intervention

Section not applicable

## 6. Study Intervention(s) and Concomitant Therapy

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

## 6.1. Study Intervention(s) Administered

In this parallel-group, randomized study, participants who meet study entry criteria will be randomly assigned in a 1:1:1 ratio to receive either 225 mg BNC210, 675 mg BNC210, or placebo.





Table 3. Study Arm(s)

| Arm Title | 225 mg BNC210 | 675 mg BNC210 | Placebo |
|---|---|---|---|
| Arm Type | Experimental | Experimental | Placebo<br>Comparator |
| Associated Intervention<br>Labels | 225 mg BNC210 | 675 mg BNC210 | Placebo |

## 6.2. Preparation/Handling/Storage/Accountability

- 1. The Investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study intervention received, and ensure any discrepancies are reported and resolved before use of the study intervention.
- 2. Only participants enrolled in the study may receive study intervention, and only authorized site staff may administer study intervention. All study intervention must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the Investigator and authorized site staff.
- 3. The Investigator, institution, or the head of the medical institution (where applicable) is responsible for study intervention accountability, reconciliation, and record maintenance (i.e., receipt, reconciliation, and final disposition records).
- 4. Further guidance and information on the handling, storage, accountability, dispensing and for the final disposition of unused study interventions are provided in the Investigational Product Manual.

## 6.3. Measures to Minimize Bias: Randomization and Blinding

#### **IWRS**

After a participant signs the ICF at Screening, site personnel will register the participant in the interactive web response system (IWRS).

Upon successful completion of the Screening Module, the system will assign the participant a unique participant number (Subject ID).

Randomization will be performed as double-blind, central randomization. The randomization schedule will be computer generated using a permuted block algorithm and will randomly allocate study intervention to randomization numbers. The randomization numbers will be assigned sequentially through the IWRS as participants enter the study. Study center will not be a blocking factor in the randomization schedule.

The randomization schedule will be prepared before the start of the study. No one involved in the study performance will have access to the randomization schedule before official unblinding of treatment assignment. No participant will be randomized into this study more than once.

Upon successful completion of randomization in the IWRS, the system will determine the correct study intervention to dispense. Once a participant is randomized to a treatment arm, the randomization will remain documented as such. The system will never reuse the same randomization number.

The system will then determine which specific wallet (with assigned number) of the assigned study intervention type is available for dispensing and inform the study site to dispense that specific wallet. The assigned wallet will correspond to the correct treatment for the participant.

# Blinding and breaking of the blind via IWRS

This is a double-blind study in which all participants, investigators, raters, and study personnel involved in the conduct of the study, including data management, will be blinded to treatment assignment, with the exception of a specified unblinded statistician and programmer who will have access to the randomization code. The unblinded study personnel will not participate in study procedures or data analysis prior to unblinding of the study data to all study-related personnel.

Study personnel will make every effort to safeguard the integrity of the study blind to minimize bias in the conduct of the study. Treatment unblinding is discouraged if knowledge of the treatment assignment will not materially change the planned management of a medical emergency. Unblinding will be permitted in a medical emergency that requires immediate knowledge of the participant's treatment assignment. Participant safety must always be the first consideration in making such a determination.

Unblinding should be discussed in advance with the Medical Monitor, if possible. If the investigator is not able to discuss treatment unblinding in advance, then they must notify the Medical Monitor as soon as possible about the unblinding incident without revealing the participant's treatment assignment.

For emergency unblinding, study personnel will use the IWRS. The IWRS will be programmed with blind-breaking instructions. If a participant's intervention assignment is unblinded, the sponsor must be notified within 24 hours of this occurrence. The date and reason that for the unblinding must be recorded.

Overall unblinding will take place at the end of the study only after database lock.

## **6.4.** Study Intervention Compliance

Study intervention will be administered at the study site under direct supervision of authorized site staff. A mouth check will be performed to ensure that the dose was swallowed.

#### 6.5. Dose Modification

Dose reductions or increases will not be allowed in this study.

## 6.6. Continued Access to Study Intervention After the End of the Study

Participants will not have access to study interventions after completion of their participation in the study. Participants should be directed to receive standard of care treatments as directed by the Investigator or their primary care physician.

#### 6.7. Treatment of Overdose

For this study, any dose of BNC210/placebo greater than 675 mg will be considered an overdose. In the event of a suspected overdose, the investigator should:

- Contact the Medical Monitor immediately.
- Closely monitor the participant for any AE/SAE and laboratory abnormalities until they have resolved or stabilized.
- Document the quantity of the excess dose.

## **6.8.** Concomitant Therapy

Any medication or vaccine (including over-the-counter or prescription medicines, recreational drugs, vitamins, and/or herbal supplements) or other specific categories of interest that the participant is receiving at the time of Screening or receives during the study must be recorded along with:

- Reason for use
- Dates of administration, including start and end dates
- Dosage information, including dose and frequency

The Medical Monitor should be contacted if there are any questions regarding concomitant or prior therapy.

Use of any investigational drug, vaccine, or invasive device within 30 days prior to Screening and at any point during the study is prohibited.

Inducers of cytochrome P450 3A4 should not be used within 30 days of Screening and their use is prohibited during the study. This includes, but is not limited to: carbamazepine, phenytoin, oxcarbazepine, barbiturates, phenobarbital, butalbital, St. John's wort, rifampicin, rifabutin, efavirenz, nevirapine, pioglitazone, troglitazone, corticosteroids by the systemic route (refer to the following website for a more extensive list <a href="https://drug-interactions.medicine.iu.edu/MainTable.aspx">https://drug-interactions.medicine.iu.edu/MainTable.aspx</a>).

Moderate to strong inhibitors of cytochrome P450 3A4 should not be used within 14 days of Screening and their use is prohibited during the study. These include grapefruit juice, verapamil, diltiazem, fluvoxamine, fluconazole and itraconazole, and HIV antivirals (refer to the following website for a more extensive list <a href="https://drug-interactions.medicine.iu.edu/MainTable.aspx">https://drug-interactions.medicine.iu.edu/MainTable.aspx</a>).

Participants who are being treated with an antidepressant medication must have discontinued the medication for at least 30 days prior to Screening (as per exclusion criterion #14) and be titrated off their medication in accordance with current prescribing guidelines. Participants must also have discontinued chronic daily use of benzodiazepines for at least 90 days prior to Screening. The withdrawal of these medications is at the discretion of the participant in consultation with their primary physician and falls outside the scope of this study protocol. Concurrent use of these medications is also prohibited during all stages of the study.

The use of any other central nervous system (CNS)-acting medications, including intermittent use of benzodiazepines, beta blockers, recreational drugs, over-the-counter medications, or herbal preparations for the treatment of symptoms of anxiety or SAD, is also not allowed within 30 days of Screening and at no time during the study.

The CNS-acting medications prohibited during the study include, but are not limited to, antidepressants, mood stabilizers, methylphenidate and other stimulants, quetiapine and other antipsychotics, anticonvulsant drugs (including gabapentinoids), zaleplon and other hypnotics, benzodiazepines, doxazosin, prazosin, clonidine, first generation sedating H1 antihistamines, zopiclone, eszopiclone, zolpidem extended-release and acetylcholinesterase inhibitors.

The use of other nonprescription medications (including herbal medications not for the treatment of symptoms of anxiety or SAD) will be discouraged during the course of the study. Prescription medications should be limited and avoided if possible, but will be allowed where clinically indicated, e.g., for treatment of AEs or pre-existing medical conditions documented at Screening.

If a medication or treatment is administered that is in breach of these restrictions, the medical monitor must be notified promptly in order to assess the participant's suitability for continued study participation.

# 7. Discontinuation of Study Intervention and Participant Discontinuation/Withdrawal

The process for discontinuation of specific sites or the study as a whole are detailed in Appendix 1: Regulatory, Ethical, and Study Oversight Considerations.

#### 7.1. Discontinuation of Study Intervention

Section not applicable.

## 7.2. Participant Discontinuation/Withdrawal from the Study

- A participant may withdraw from the study at any time at his/her own request or may be
  withdrawn at any time at the discretion of the Investigator for safety, behavioral, or
  compliance reasons. This is expected to be uncommon.
- If the participant had received study intervention prior to discontinuing from the study, a Follow-up Visit should be conducted if possible, as shown in the SoA (Section 1.3).
- If the participant withdraws consent for disclosure of future information, the Sponsor may retain and continue to use any data collected before such a withdrawal of consent.
- If a participant withdraws from the study, he/she may request destruction of any samples taken and not tested, and the Investigator must document this in the site study records.

## 7.3. Lost to Follow-up

A participant will be considered lost to follow-up if he/she repeatedly is unable to be contacted by the study site for the Follow-up Visit.

The following actions must be taken if a participant initially is unable to be contacted for the Follow-up Visit:

- The site must attempt to contact the participant and reschedule the missed visit/appointment as soon as possible and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

## 8. Study Assessments and Procedures

- Study procedures and their timing are summarized in the SoA (Sections 1.3 and 1.4). Protocol waivers or exemptions are not allowed.
- Immediate safety concerns should be discussed with the Medical Monitor immediately upon occurrence or awareness to determine if the participant should continue on study.
- Adherence to the study design requirements, including those specified in the SoA (Sections 1.3 and 1.4), is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The Investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.



- At the conclusion of the post-challenge assessment period on the Treatment Day, the Investigator should assess the participant's suitability to be discharged from the study site based on their medical judgment.
- Visits scheduled due to increased safety monitoring, if applicable, must be captured as an unscheduled visit. All assessments completed during an unscheduled visit must be captured in the electronic case report form (eCRF). This includes the results of all pathology tests scheduled by the Investigator.
- A visit with a participant's primary physician (i.e., not a study Investigator) is not considered an unscheduled visit. Similarly, hospital admissions due to SAEs are also not considered unscheduled visits. Assessments completed by external institutions should not be entered into the eCRF.
## 8.1. Efficacy Assessments

Planned timepoints for all efficacy assessments are provided in the SoA (Section 1.3 and 1.4).



## 8.1.2. Subjective Units of Distress Scale (SUDS)

The SUDS measures the subjective intensity of disturbance or distress currently experienced by an individual and is a standard instrument for rating social and performance anxiety in patients with SAD during role-playing situations. The individual self-assesses where they are on the scale, between 0-100, with higher numbers indicating more anxiety/greater discomfort (Wolpe, 1969, Heimberg 1998, 2002).

#### 8.1.3. Spielberger State-Trait Anxiety Inventory (STAI)

The STAI (<u>Spielberger 1983</u>) is a widely used self-report measure of subjective anxiety in clinical practice. It comprises 2 scales of 20 items asking participants to report their feelings of anxiousness: the STAI-State scale requires reporting of feelings at the time of questionnaire completion and the STAI-Trait scale requires reporting of how the subject generally feels. Responses are marked on a 4-point scale from "not at all" to "very much so." The STAI-State component only will be used in this study.

#### 8.1.4. Self-Statements During Public Speaking (SSPS)

The SSPS is a self-report instrument that assesses cognitions related to public speaking (Hofmann 2000). The original version of the SSPS assesses how a participant typically thinks/feels during any public speaking situation (SSPS-Trait). The SSPS has also been modified and validated to assess how a participant feels at the time of questionnaire completion in relation to a current public speaking situation (SSPS-State) (Osorio 2013). Both the SSPS-Trait and SSPS-State versions will be used in this study at the time points specified in Section 1.4. The SSPS is a 10-item questionnaire consisting of two 5-item subscales, the Positive Self-Statements (SSPS-P) and the Negative Self-Statements (SSPS-N). Only the SSPS-N subscale will be included in the secondary endpoint analyses in this study.

## 8.2. Safety Assessments

Planned timepoints for all safety assessments are provided in the SoA (Section 1.3).

## 8.2.1. Physical Examinations

- A complete physical examination will include, at a minimum, assessments of the general appearance, skin and lymphatics, eyes, ears, nose, throat, cardiovascular system, respiratory system, abdomen/gastrointestinal system, musculoskeletal, and neurological systems. Other body systems may also be examined as required. Height and weight will also be measured at Screening only.
- An abbreviated physical examination will include, at a minimum, assessments of the eyes, ears, nose, throat, cardiovascular system, respiratory system, and abdomen/gastrointestinal system. Other body systems may also be examined as required.

#### 8.2.2. Vital Signs

- Body temperature, pulse rate, respiratory rate, and systolic and diastolic blood pressure will be assessed.
- Blood pressure and pulse measurements will be assessed in a seated position with a completely automated device. Manual techniques will be used only if an automated device is not available.
- Blood pressure and pulse measurements should be preceded by at least 5 minutes of rest in a seated position for the participant in a quiet setting without distractions (e.g., television, cell phones).

#### 8.2.3. Electrocardiograms

- Triplicate 12-lead ECGs will be obtained as outlined in the SoA (Section 1.3) using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
- At each time point, 3 individual ECG tracings should be obtained in succession, approximately 2 minutes apart.
- One repeat is allowed for screening purposes if abnormal findings are observed. The repeat must also be completed in triplicate.
- Participants must be resting in a semi-supine or supine position for at least 5 minutes prior to obtaining ECG.
- The same ECG machine should be used for all recordings from an individual participant, where possible.
- ECGs will be read by the Investigator or designated physician.
- QTcF values will be derived from the data available and the average QTcF will be used when assessing eligibility.

For safety monitoring purposes, the Investigator or designee must review, sign, and date all ECG tracings. Paper copies will be kept at the study center with the participant's clinical file as part of the permanent record. The ECG intervals and interpretation will be recorded on the appropriate eCRF.

Paper ECG recordings should be photocopied and maintained as a permanent source document. The Sponsor reserves the right to request copies of paper ECG recordings for independent cardiology review.

#### 8.2.4. Clinical Safety Laboratory Assessments

- See Appendix 2: Clinical Laboratory Tests for the list of clinical laboratory tests to be performed and to the SoA (Section 1.3) for the timing and frequency.
- The Investigator must review the laboratory report, document this review, and record any
  clinically significant changes occurring during the study as an AE. The laboratory reports
  must be filed with the source documents.
- All laboratory tests with values considered clinically significantly abnormal during
  participation in the study should be repeated until the values return to normal or baseline
  or are no longer considered clinically significant by the Investigator or Medical Monitor.
  - If clinically significant values do not return to normal/baseline within a period of time judged reasonable by the Investigator, the etiology should be identified, and the medical monitor/sponsor notified.
  - All protocol-required laboratory tests, as defined in Appendix 2: Clinical Laboratory Tests, must be conducted in accordance with the Laboratory Manual and the SoA (Section 1.3).
  - If laboratory values from non-protocol specified laboratory tests performed at the institution's local laboratory require a change in participant management or are considered clinically significant by the investigator (e.g., SAE or AE), then the results must be recorded.
  - All events of ALT or AST ≥3 × ULN and total bilirubin ≥2 × ULN (>35% direct bilirubin) which may indicate severe liver injury (possible Hy's Law), as well as all events of ALT or AST ≥ 5 x ULN, must be reported to the medical monitor in an expedited manner. Details of required actions and follow-up are given in Appendix 5: Liver Safety: Suggested Actions and Follow-up Assessments.

#### 8.2.5. Suicidal Ideation and Behavior Risk Monitoring

BNC210 is considered to be a CNS-active intervention.

Baseline assessment of suicidal ideation and behavior will be assessed using the C-SSRS.

The C-SSRS is a suicidal ideation rating scale designed to identify behaviors that may be indicative of a participant's intent to commit suicide. The scale is administered via a semi-structured interview and measures both passive and active suicidal ideation and the intensity and duration of the ideation. Both suicidal and non-suicidal self-injurious behavior is also assessed.

Prior to the participant being discharged from the study site on the Treatment Day, the Investigator will assess any intervention-emergent suicidal behavior as part of their overall assessment of the participant's suitability to be discharged.

## 8.3. Adverse Events (AEs), Serious Adverse Events (SAEs), and Other Safety Reporting

The definitions of AEs and SAEs can be found in Appendix 3: AEs and SAEs: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting.

AEs will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).

The Investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible for following up all AEs/SAEs.

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 3: AEs and SAEs: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting.

## 8.3.1. Time Period and Frequency for Collecting AE and SAE Information

All SAEs will be collected from the signing of the ICF until the Follow-up Visit at the timepoints specified in the SoA (Section 1.3).

All AEs will be collected from the start of intervention until the Follow-up Visit at the timepoints specified in the SoA (Section 1.3). Medical occurrences that begin before the start of study intervention, but after obtaining informed consent will be recorded as medical history/current medical conditions, not as AEs.

All SAEs will be recorded and reported to the sponsor or designee immediately and under no circumstance should this exceed 24 hours, as indicated in Appendix 3: AEs and SAEs: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting. The Investigator will submit any updated SAE data to the Sponsor within 24 hours of it being available.

Investigators are not obligated to actively seek information on AEs or SAEs after conclusion of the study participation. However, if the Investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study intervention or study participation, the Investigator must promptly notify the Sponsor.

#### 8.3.2. Method of Detecting AEs and SAEs

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the participant is the preferred method to inquire about AE occurrences.

#### 8.3.3. Follow-up of AEs and SAEs

After the initial AE/SAE report, the Investigator is required to proactively follow each participant at subsequent visits/contacts. All SAEs will be followed until resolution, stabilization, the event is otherwise explained, or the participant is lost to follow-up (as defined in Section 7.3). Further information on follow-up procedures is provided in Appendix 3: AEs and SAEs: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting.

#### 8.3.4. Regulatory Reporting Requirements for SAEs

- Prompt notification by the Investigator to the Sponsor of an SAE is essential so that legal
  obligations and ethical responsibilities to the safety of participants and the safety of a
  study intervention under clinical investigation are met.
- The Sponsor has a legal responsibility to notify both the local regulatory authority and
  other regulatory agencies about the safety of a study intervention under clinical
  investigation. The Sponsor will comply with country-specific regulatory requirements
  relating to safety reporting to the regulatory authority, Institutional Review Board (IRB)
  and Investigators.
- An Investigator who receives an investigator safety report describing an SAE or other specific safety information (e.g., summary or listing of SAEs) from the Sponsor will review and then file it along with the IB and will notify the IRB, if appropriate according to local requirements.

## 8.3.5. Pregnancy

- Details of all pregnancies in female participants and female partners of male participants w
  ill be collected after the start of study intervention and until 1 week after the last dose of
  study intervention is administered.
- If a pregnancy is reported in a female participant or female partner of male participant (after obtaining the necessary signed informed consent from the female partner), the Investigator will record pregnancy information on the appropriate form and submit it promptly, within 24 hours of learning of the pregnancy, signing and dating the Pregnancy Data Collection Form, verifying the accuracy of the information recorded in the form with the source documents and eCRF. Pregnancy reporting contact information can be found in Appendix 3, Section 10.3.4.
- While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy for medical reasons will be reported as an AE or SAE.
- Abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs and will be reported as such.
- The participant/pregnant female partner will be followed to determine the outcome of the pregnancy. The Investigator will collect follow-up information on the participant/pregnant female partner and the neonate and the information will be forwarded to the Sponsor.

- Any post-study pregnancy-related SAE considered reasonably related to the study intervention by the Investigator will be reported to the Sponsor as described in Section 8.3.4. While the Investigator is not obligated to actively seek this information in former study participants/pregnant female partner, he or she may learn of an SAE through spontaneous reporting.
- Any female participant who becomes pregnant while participating in the study will discontinue study intervention and be withdrawn from the study.

## 8.4. Plasma Bioanalysis

- Whole blood samples of approximately 4 mL will be collected for measurement of plasma concentrations of BNC210 as specified in the SoA (Section 1.3).
- As the study is double-blind, samples will be collected from all participants, but only those allocated to BNC210 treatment arms will have their samples analyzed.
- Instructions for the collection and handling of biological samples will be provided by the Sponsor in the study-specific Laboratory Manual.

#### 8.5. Genetics

Genetics are not evaluated in this study.

#### 8.6. Biomarkers

Biomarkers are not evaluated in this study.

## 8.7. Immunogenicity Assessments

Not applicable.

#### **8.8.** Medical Resource Utilization and Health Economics

Medical resource utilization and health economics parameters are not evaluated in this study.

#### 9. Statistical Considerations

The statistical analysis plan (SAP) will be finalized prior to database lock and it will include a more technical and detailed description of the statistical analyses described in this section. This section is a summary of the planned statistical analyses of the most important endpoints, including primary and secondary endpoints.

## 9.1. Statistical Efficacy Hypotheses

The primary objective of this study is to assess the effects of a single dose of BNC210 compared to placebo on change in self-reported anxiety severity as measured by the SUDS from baseline to the performance phase in a public speaking challenge.

• The null hypothesis for the primary efficacy endpoint of equality of a single dose of BNC210 and placebo is:

H<sub>01</sub>: Mean changes in SUDS scores between baseline and the average of the performance phase in a public speaking challenge between either single dose (225 mg or 675 mg) of BNC210 and placebo are equal

To assess the effects of BNC210 compared to placebo in reducing self-reported anxiety

The secondary objectives of this study and their respective null hypotheses of the equality of a single dose (225 mg or 675 mg) of BNC210 and placebo are:

severity as measured by the SUDS in a public speaking challenge

| H <sub>02</sub> : Mean changes in SUDS scores between baseline and the average of t phase in a public speaking challenge between either single dose (225 mg of BNC210 and placebo are equal |
|---|

- To assess the effects of BNC210 compared to placebo in reducing self-reported symptoms of anxiety as measured by the STAI-State in a public speaking challenge
  - H<sub>06</sub>: Mean changes in STAI-State scores between baseline and the performance phase in a public speaking challenge between either single dose (225 mg or 675 mg) of BNC210 and placebo are equal
  - H<sub>07</sub>: Mean changes in STAI-State scores between baseline and the anticipation phase in a public speaking challenge between either single dose (225 mg or 675 mg) of BNC210 and placebo are equal
- To assess the effects of BNC210 compared to placebo in reducing self-reported negative cognitions during speaking as measured by the SSPS-N in a public speaking challenge

H<sub>08</sub>: Mean changes in SSPS-N scores between baseline and the performance phase in a public speaking challenge between either single dose (225 mg or 675 mg) of BNC210 and placebo are equal

H<sub>09</sub>: Mean changes in SSPS-N scores between baseline and the anticipation phase in a public speaking challenge between either single dose (225 mg or 675 mg) of BNC210 and placebo are equal

#### 9.1.1. Multiplicity Adjustment

Because this is a Phase 2 study, the level of significance will be set at 0.05 for primary and secondary endpoints with no adjustment for multiple comparisons.

## 9.2. Analysis Sets

The following analysis populations are planned for this study:

- Safety Population (SAF): The safety population includes all participants who receive any amount of the study intervention. The safety population will be used for the analysis of the safety endpoints. Participants will be analyzed by actual treatment received.
- Intent-to-Treat Population (ITT): The ITT population includes all randomized participants. Participants will be analyzed by randomized treatments.
- Full Analysis Set (FAS): The FAS population includes all participants in the ITT population who receive any amount of the study intervention. Participants will be analyzed by randomized treatment.

| Per-Protocol Population (PP): The FAS population who have no | he per-protocol population will include participants |
|---|---|
| ine 1745 population who have no | major protocor deviations. |
| | Participants will be analyzed by |
| randomized treatments. | r articipants will be analyzed by |

## 9.3. Statistical Analyses

#### 9.3.1. General Considerations

This section presents a summary of the planned statistical analyses. A SAP that describes the details of the analyses to be conducted will be written prior to the study database being locked.

Unless otherwise indicated, all testing of statistical significance will be two-sided and a difference resulting in a p value of  $\leq 0.05$  will be considered statistically significant.

Summary statistics will be provided for the variables described below. For continuous variables, these statistics will typically include the number of participants, mean, standard deviation (SD), median, minimum, and maximum. For categorical variables, these statistics will typically include the number and percentage of participants in each category.

## 9.3.2. Study Participants and Demographics

#### 9.3.2.1. Disposition and Withdrawals

The number of participants randomized, completing, and withdrawing, along with reasons for withdrawal, will be tabulated overall and by treatment group. The number of participants in each analysis population will be reported.

#### 9.3.2.2. Protocol Deviations

Protocol deviations will be identified and classified as important or non-important for statistical analysis purposes before unblinding and will be summarized or listed as appropriate. Important protocol deviations that might affect efficacy data will be used to exclude participants from the per-protocol analysis.

#### 9.3.2.3. Demographics and Other Baseline Characteristics

The following analyses will be conducted for all analysis populations:

- Demographic variables will include age, sex, height, and weight. Information on race and ethnicity will be collected for any eventual analysis of differences in response to the study intervention in accordance with local regulatory requirements. Baseline participant characteristics will include whether the participant wore a mask during the performance phase of the public speaking challenge, medical history, including confirmation of SAD diagnosis, and LSAS total score at Screening. Baseline evaluation of the SUDS score, STAI-State score, and SPSS-N score will also be reported.
- Prior and concomitant medications will be summarized by treatment group, by the number and percentage of participants taking each medication, classified using World Health Organization Drug Dictionary (WHO-DD) Anatomical Therapeutic Chemical (ATC) classes and preferred terms.

#### 9.3.3. Primary Endpoint(s)/Estimand(s) Analysis

The primary efficacy endpoint for the current study will be the difference in change in SUDS sc ores after oral administration of a single dose of BNC210 and placebo. The analysis of the primary efficacy endpoint will be evaluated for the FAS and PP populations according to the planned treatment.

The primary endpoint will be assessed with a longitudinal linear mixed-effects model for each SUDS timepoint, with the average of each timepoint in the performance phase used as the final timepoint. The model will include fixed effects for treatment, interaction between treatment and timepoint, sex, mask usage and a covariate for baseline score. Baseline will be defined in detail in the SAP.

Two comparisons (BNC210 225 mg versus placebo and BNC210 675 mg versus placebo) will be made and the least squares (LS) mean difference along with the corresponding 95% confidence interval (CI) will be reported. For each treatment arm, the LS mean difference along with the corresponding *p* value will be weighted equally across the 2 BNC210 arms.

| 9.3.4. | Secondary Endpoints Analysis |
|---|---|
| ly the FA | cherwise specified, continuous secondary endpoints will be analyzed on or as population using a longitudinal linear mixed-effects model for each timepoint, as a for the primary analysis. |
| score of to | Additionally, the average the SUDS will be analyzed for the anticipation endpoints. STAI-State scores and SSPS-N scores will also zed as measured for the performance, anticipation, |
| <b>9.4.</b> No interi | Interim Analysis m analysis is planned for this study. |

## 10. Supporting Documentation and Operational Considerations

## 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

## 10.1.1. Regulatory and Ethical Considerations

- This study will be conducted in accordance with the protocol and with the following:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines
  - Applicable International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guidelines
  - Applicable laws and regulations
- The protocol, protocol amendments, ICF, IB, and other relevant documents (e.g., advertisements) must be submitted to an IRB by the Investigator and reviewed and approved by the IRB before the study is initiated.
- The protocol cannot be altered or changed except through a formal protocol amendment, which requires written approval from the Sponsor. Any amendments to the protocol will require IRB approval and health authority approval, where applicable, and must be signed by the Investigator before implementation of changes, except for changes necessary to eliminate an immediate hazard to study participants.
- The Investigator will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB
  - Notifying the IRB of SAEs or other significant safety findings as required by IRB procedures
  - o Providing oversight of the conduct of the study at the site and adherence to requirements of 21 CFR, ICH guidelines, the IRB, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations

#### 10.1.2. Financial Disclosure

Investigators and Sub-Investigators will provide the Sponsor with sufficient, accurate financial information as requested to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### 10.1.3. Informed Consent Process

- The Investigator or his/her representative will explain the nature of the study, including the risks and benefits, to the participant and answer all questions regarding the study.
- Participants must be informed that their participation is voluntary. Participants will be required to sign a statement of informed consent that meets the requirements of 21 CFR 50, local regulations, ICH guidelines, privacy and data protection requirements, where applicable, and the IRB or study center.
- The rights and welfare of the participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Participants must be reconsented to the most current version of the ICF(s) during their participation in the study.
- A copy of the ICF(s) must be provided to the participant.
- Informed consent will be obtained before the participant can participate in the study.
- The Investigator or his/her representative must also explain to the participant that they are completely free to refuse to enter the study or to withdraw from it at any time.
- Participants who are rescreened are required to sign a new ICF.
- Participants who are rescreened will not need to repeat routine clinical laboratory
  assessments or ECGs if an eligible result from the prior screening period has been
  obtained within 14 days of randomization into the study.
- The ICF will contain a separate section that addresses the use of remaining mandatory samples for optional exploratory research.

#### 10.1.4. Data Protection

- Participants will be assigned a unique identifier as part of their study participation. Any
  participant records or datasets that are transferred to the Sponsor will contain the
  identifier and information collected as part of the study only; participant names or any
  information that would make the participant identifiable will not be transferred.
- The participant must be informed that his/her personal study-related data will be used by the Sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant, who will be required to give consent for their data to be used as described in the ICF.
- The study data entry and study management systems used by clinical sites and by the Sponsor/designee will be secured and password protected.
- The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB members, and by inspectors from regulatory authorities.

#### 10.1.5. Data Quality Assurance

- All participant data relating to the study will be recorded in the eCRF unless transmitted to the Sponsor or designee electronically (e.g., laboratory data). The Investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the eCRF.
- Guidance on completion of eCRFs will be provided in the study-specific eCRF completion guidelines.
- The Investigator must permit study-related monitoring, audits, IRB review, and regulatory agency inspections and provide direct access to source data documents.
- Quality tolerance limits (QTLs) will be predefined in the study-specific Risk Log to
  identify systematic issues that can impact participant safety and/or reliability of study
  results. These predefined parameters will be monitored during the study, and important
  deviations from the QTLs and remedial actions taken will be summarized in the Clinical
  Study Report.
- Monitoring details describing strategy, including definition of study critical data items
  and processes (e.g., risk-based initiatives in operations and quality such as risk
  management and mitigation strategies and analytical risk-based monitoring), methods,
  responsibilities, and requirements, including handling of noncompliance issues and
  monitoring techniques (central, remote, or on-site monitoring) are provided in the
  Clinical Monitoring Plan.
- The Sponsor or designee is responsible for the data management of this study, including quality checking of the data.
- The Sponsor assumes accountability for actions delegated to other individuals (e.g., contract research organizations).
- Records and documents, including signed ICFs, pertaining to the conduct of this study
  must be retained by the Investigator for 15 years after study completion unless local
  regulations or institutional policies require a longer retention period. No records may be
  destroyed during the retention period without the written approval of the Sponsor. No
  records may be transferred to another location or party without written notification to the
  Sponsor.

#### 10.1.6. Source Documents

- Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the Investigator's site.
- Data entered in the eCRF that are transcribed from source documents must be consistent with the source documents, or the discrepancies must be explained. The Investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.

- Examples of acceptable source documentation include, but are not limited to, hospital records, clinic and office charts, laboratory notes, recorded data from automated instruments, memoranda, and pharmacy dispensing records. The Investigator must maintain accurate documentation (source data) that supports the information entered in the eCRF.
- Study monitors will perform ongoing source data verification to confirm that data entered into the eCRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.

#### 10.1.7. Study and Site Closure

The Sponsor or designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the Sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The Investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the Sponsor or investigator may include, but are not limited to:

For study termination:

• Discontinuation of further study intervention development

For site termination:

- Failure of the Investigator to comply with the protocol, the requirements of the IRB or local health authorities, the Sponsor's procedures, or GCP guidelines
- Inadequate or no recruitment (evaluated after a reasonable amount of time) of participants by the Investigator
- Total number of participants included earlier than expected

If the study is prematurely terminated or suspended, the Sponsor shall promptly inform the Investigators, the IRBs, the regulatory authorities, and any contract research organization(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements. The Investigator shall promptly inform the participant and should assure appropriate participant therapy and/or follow-up.

#### 10.1.8. Publication Policy

The publication policy is outlined in the study site-specific Clinical Trial Agreement.

## 10.2. Appendix 2: Clinical Laboratory Tests

- The tests detailed in Table 4 will be performed by the central laboratory at the timepoints described in the SoA (Section 1.3).
- Local laboratory results may only be required in the event that the central laboratory
  results are not available in time to support urgent safety or study intervention
  administration decisions, following consultation with the Medical Monitor. If a local
  sample is required, it is important that the sample for central analysis is also obtained,
  where possible. Additionally, if the local laboratory results are used to make either a
  study intervention decision or response evaluation, the results must be recorded.
- Protocol-specific requirements for inclusion or exclusion of participants are detailed in Section 5 of the protocol.
- Additional tests may be performed at any time during the study as determined necessary by the Investigator or required by local regulations.

Table 4. Protocol-Required Safety Laboratory Tests

| Laboratory<br>Tests | | | Parameters | |
|---|---|---|---|---|
| Hematology | Platelet Count | | RBC Indices: | White blood cell |
| | Red blood cell (RBC) Count Hemoglobin Hematocrit | | MCV<br>MCH<br>%Reticulocytes | (WBC) count<br>with Differential: |
| | | | | Neutrophils |
| | | | | Lymphocytes |
| | | | | Monocytes |
| | | | | Eosinophils |
| | | | | Basophils |
| Clinical | Blood urea | Potassium | Aspartate Transaminase | Total and direct |
| Chemistry <sup>1</sup> | nitrogen (BUN) | | (AST) | bilirubin |
| | Creatinine | Sodium | Alanine Transaminase | Total protein |
| | | | (ALT | |
| | Glucose | Calcium | Alkaline phosphatase <sup>2</sup> | |
| Routine<br>Urinalysis | | | inogen, pH, glucose, protein, b<br>cyte esterase, color, appearance | |
| | Microscopic examination (if blood or protein is abnormal) | | | |
| Pregnancy<br>testing | Highly sensitive serum human chorionic gonadotropin (hCG) pregnancy test (as needed for women of childbearing potential) <sup>3</sup> | | | |

| Laboratory<br>Tests | Parameters |
|---|---|
| Other | Urine drug test at Screening |
| Screening<br>Tests | <ul> <li>Follicle-stimulating hormone and estradiol (as needed in women of<br/>non-childbearing potential only)</li> </ul> |
| | <ul> <li>Serology (HIV antibody, hepatitis B surface antigen [HBsAg], and<br/>hepatitis C virus antibody)</li> </ul> |
| | <ul> <li>All study-required laboratory tests will be performed by a central<br/>laboratory, with the exception of:</li> </ul> |
| | Urine drug test at Baseline / Pre-dose |
| | <ul> <li>Urine pregnancy test at Baseline / Pre-dose<sup>3</sup></li> </ul> |

#### NOTES:

- 1. All events of ALT or AST  $\geq 3 \times$  upper limit of normal (ULN) and total bilirubin  $\geq 2 \times$  ULN (>35% direct bilirubin), which may indicate severe liver injury (possible Hy's Law), as well as all events of ALT or AST  $\geq 5 \times$  ULN, must be reported to the Medical Monitor in an expedited manner. Details of required actions and follow-up are given in Appendix 5: Liver Safety: Suggested Actions and Follow-up Assessments.
- 2. If alkaline phosphatase is elevated, consider fractionating.
- 3. Local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB.

Abbreviations: HIV = human immunodeficiency virus; MCH = mean corpuscular hemoglobin; MCV = mean corpuscular volume

Investigators must document their review of each laboratory safety report.

## 10.3. Appendix 3: AEs and SAEs: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### 10.3.1. Definition of AE

#### **AE Definition**

- An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.

#### Definition of Unsolicited and Solicited AE

- An unsolicited AE is an AE that was not solicited using a Participant Diary and that is communicated by a participant who has signed the informed consent. Unsolicited AEs include serious and non-serious AEs.
- Potential unsolicited AEs may be medically attended (i.e., symptoms or illnesses
  requiring a hospitalization, or emergency room visit, or visit to/by a health care
  provider). The participant will be instructed to contact the site as soon as possible to
  report medically attended event(s), as well as any events that, though not medically
  attended, are of participant concern. Detailed information about reported unsolicited
  AEs will be collected by qualified site personnel and documented in the participant's
  records.
- Unsolicited AEs that are not medically attended nor perceived as a concern by a
  participant will be collected during interview with the participant and by review of
  available medical records at the next visit.
- Solicited AEs are predefined local and systemic events for which the participant is specifically questioned, and which are noted by the participant.

#### **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or
  other safety assessments (e.g., ECG, radiological scans, vital signs measurements),
  including those that worsen from baseline, considered clinically significant in the
  medical and scientific judgment of the Investigator (i.e., not related to progression of
  underlying disease).
- Exacerbation of a chronic or intermittent pre-existing condition, including either an increase in frequency and/or intensity of the condition.

- New conditions detected or diagnosed after study intervention administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected intervention-intervention interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study
  intervention or a concomitant medication. Overdose per se will not be reported as an
  AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming
  intent. Such overdoses should be reported regardless of sequelae.
- The signs, symptoms, and/or clinical sequelae resulting from lack of efficacy will be reported as AE or SAE if they fulfil the definition of an AE or SAE. "Lack of efficacy" or "failure of expected pharmacological action" also constitutes an AE or SAE.

## **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety
  assessments that are associated with the underlying disease, unless judged by the
  Investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (e.g., endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 10.3.2. Definition of SAE

An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed:

#### a. Results in death

#### b. Is life threatening

The term *life threatening* in the definition of *serious* refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

#### c. Requires inpatient hospitalization or prolongation of existing hospitalization

• In general, hospitalization signifies that the participant has been admitted (usually involving at least an overnight stay) at the hospital or emergency ward for observation

and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether hospitalization occurred or was necessary, the AE should be considered serious.

 Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

### d. Results in persistent or significant disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle) that may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### e. Is a congenital anomaly/birth defect

#### f. Other Important Medical Event:

- Medical or scientific judgment should be exercised by the Investigator in deciding
  whether SAE reporting is appropriate in other situations, such as significant medical
  events that may jeopardize the participant or may require medical or surgical
  intervention to prevent one of the other outcomes listed in the above definition. These
  events should usually be considered serious.
  - Examples of such events include invasive or malignant cancers, intensive treatment for allergic bronchospasm, blood dyscrasias, convulsions, or development of intervention dependency or intervention abuse.

#### 10.3.3. Recording and Follow-Up of AE and/or SAE

#### AE and SAE Recording

The Investigator is responsible for the detection and documentation of events meeting the criteria and definition of an AE or SAE described previously.

- At each specified time point, the participant will be allowed time to spontaneously report any issues since the last visit or evaluation. The Investigator will then monitor and/or ask about or evaluate AEs using non-leading questions, such as
  - o "How are you feeling?"
  - o "Have you experienced any issues since your last visit?"
  - o "Have you taken any new medications since your last visit?"
- Any clinically relevant observations made during the visit will also be considered AEs.

- When an AE/SAE occurs, it is the responsibility of the Investigator to review all
  documentation (e.g., hospital progress notes, laboratory reports, and diagnostics
  reports) related to the event.
- The Investigator will then record all relevant AE/SAE information.
- It is **not** acceptable for the Investigator to send photocopies of the participant's medical records to the Sponsor or designee in lieu of completion of the required form.
- There may be instances when copies of medical records for certain cases are requested
  by the Sponsor or designee. In this case, all participant identifiers, with the exception
  of the participant number (Subject ID), will be redacted on the copies of the medical
  records before submission to the Sponsor or designee.
- The Investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

#### Assessment of Intensity

The Investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to one of the following categories:

- Mild: Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
- Moderate: Minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental Activities of Daily Living (ADL). Instrumental ADL refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
- Severe: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling, limiting self-care ADL. Self-care ADL refers to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

#### **Assessment of Causality**

The Investigator is obligated to assess the relationship between study intervention and each occurrence of each AE/SAE.

- The Investigator will also consult the IB and/or product information, for marketed products, in his/her assessment.
- For each AE/SAE, the Investigator **must** document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.

- There may be situations in which an SAE has occurred, and the Investigator has
  minimal information to include in the initial report to the Sponsor or designee.
  However, it is very important that the Investigator always make an assessment of
  causality for every event before the initial transmission of the SAE data to the Sponsor
  or designee.
- The Investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.

The causality assessment is one of the criteria used when determining regulatory reporting requirements.

The Investigator will use clinical judgment to determine the relationship following the below definitions:

- Not Related: This category applies to an AE that is clearly not related to the
  investigational agent/procedure, beyond a reasonable doubt. That is, another cause of
  the event is most plausible; and/or a clinically plausible temporal sequence is
  inconsistent with the onset of the event and the administration of study intervention
  and/or a causal relationship is considered biologically implausible.
- Unlikely Related: This category applies to an AE that could reasonably be considered
  caused by something else, and where there is no known or expected response pattern to
  the suspected study intervention.
- Possibly Related: This category applies to an AE that follows a reasonable temporal
  sequence from administration of the study intervention and that follows a known or
  expected response pattern to the suspected study intervention, but that could readily
  have been produced by a number of other factors
- Probably Related: This category applies to an AE that follows a reasonable temporal
  sequence from administration of the study intervention; that follows a known response
  pattern to the suspected study intervention; that is confirmed by an improvement on
  stopping the study intervention; and that cannot be reasonably explained by the
  participant's clinical state.
- Definitely Related: This category applies to an AE that is plausible, and concurrent
  disease or other drugs or chemicals cannot explain event. The response to withdrawal
  of the study intervention (dechallenge) should be clinically plausible. The event must
  be definitive pharmacologically or phenomenologically, using a satisfactory
  rechallenge procedure if necessary.

## Follow-up of AEs and SAEs

• The Investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by the Sponsor or designee to elucidate the nature and/or causality of the AE or SAE as fully as

possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.

- If a participant dies during participation in the study or during a recognized follow-up period, the Investigator will provide the Sponsor or designee with a copy of any postmortem findings including histopathology, if available and appropriate.
- New or updated information will be recorded using a new copy of the SAE Report
  Form and contain the site and Investigator information, participant information, SAE,
  and SAE onset date as minimum reporting information, as well as all new information
  and all data changed. It should be made clear whether the new information is in
  addition to or meant to replace the previously reported information.
- The Investigator will submit any updated SAE data to the Sponsor or designee within 24 hours of receipt of the information.

## 10.3.4. Reporting of SAEs

| SAE Reporting |
|---|
| The Investigator or designee must report all SAEs promptly |
| within 24 hours of first becoming aware of the event by |
| completing, signing, and dating the SAE Report Form, verifying the accuracy of the information recorded in the form with the source documents and eCRF, and sending the SAE |
| Report Form by one of the following |
| methods: |
| THE SECOND SECON |

This written report should be submitted on the SAE form provided for this purpose. At the time of first notification, the Investigator or designee should provide the following information, if available:

- Protocol number
- Reporter (study site and Investigator)
- Participant number (Subject ID)
- Participant's year of birth
- Participant's sex
- Date of study intervention dose
- Date of last dose of study intervention prior to SAE onset, if applicable
- SAE term
- Date of occurrence of the event

- Severity of the SAE term
- A brief description of the event, treatment, outcome to date, and any actions taken with study intervention
- The seriousness criteria(on) that were met
- Investigator causality assessment
- Concomitant medications taken within 30 days of onset of the event
- Relevant medical history information
- Relevant laboratory test findings
- Whether and when the Investigator was unblinded as to the participant's treatment assignment

Any missing or additional relevant follow-up information concerning the SAE should be sent via the same contact details above as soon as possible on a follow-up SAE Report Form, together with the following minimal information: initial report, AE, date of occurrence, study participant identifier, and site number. This will allow the follow-up information to be linked to the initial SAE report.

Specific information may be requested by

using a follow-up request form or via email communication.

The Investigator is required to comply with applicable regulations (including local laws and guidances) regarding the notification of his or her health authorities, IRB, principal and coordinating investigators, study investigators, and institutions. Each Investigator is obligated to learn about the reporting requirements for investigators in his/her country. The study monitor may be able to assist with this.

## 10.4. Appendix 4: Contraceptive and Barrier Guidance

#### 10.4.1. Definitions

## Woman of Childbearing Potential (WOCBP)

Women in the following categories are considered WOCBP (fertile):

- 1. Following menarche
- 2. From the time of menarche until becoming postmenopausal unless permanently sterile (see below)
- A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
  - A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, confirmation with more than one FSH measurement and FSH levels within the institutional postmenopausal range is required.
  - o Females on HRT and whose menopausal status is in doubt will be required to use one of the nonestrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.
- Permanent sterilization methods (for the purpose of this study) include:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy
  - For individuals with permanent infertility due to an alternate medical cause other than the above, (e.g., Mullerian agenesis, androgen insensitivity, gonadal dysgenesis), investigator discretion should be applied to determining study entry.

**Note:** Documentation can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.

 If fertility is unclear (e.g., amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before first dose of study intervention, additional evaluation should be considered.

#### 10.4.2. Contraception Guidance

#### CONTRACEPTIVES<sup>a</sup> ALLOWED DURING THE STUDY INCLUDE:

#### Highly Effective Methods<sup>b</sup> That Have Low User Dependency

- Implantable progestogen-only hormone contraception associated with inhibition of ovulation<sup>c</sup>
- Intrauterine device (IUD)
- Intrauterine hormone-releasing system (IUS)<sup>c</sup>
- Bilateral tubal occlusion
- Azoospermic partner (vasectomized or due to a medical cause)

Azoospermia is a highly effective contraceptive method provided that the partner is the sole sexual partner of the woman of childbearing potential and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used. Spermatogenesis cycle is approximately 90 days. Note: documentation of azoospermia for a male participant can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.

#### Highly Effective Methods<sup>b</sup> That Are User Dependent

- Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation<sup>c</sup>
  - o oral
  - o intravaginal
  - o transdermal
  - o injectable
- Progestogen-only hormone contraception associated with inhibition of ovulation<sup>c</sup>
  - oral
  - o injectable
- Sexual abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

- a) Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for those participating in clinical studies.
- b) Failure rate of < 1% per year when used consistently and correctly. Typical use failure rates differ from those when used consistently and correctly.
- c) Male condoms must be used in addition to hormonal contraception. If locally required, in accordance with Clinical Trial Facilitation Group (CTFG) guidelines, acceptable contraceptive methods are limited to those which inhibit ovulation as the primary mode of action.

Note: Periodic abstinence (calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method (LAM) are not acceptable methods of contraception for this study. Male condom and female condom should not be used together (due to risk of failure from friction).

# 10.5. Appendix 5: Liver Safety: Suggested Actions and Follow-up Assessments

The table below describes suggested actions and follow-up assessments should a participant's post-challenge clinical safety laboratory results meet the following criteria.

| ost-chancinge chinical sa | icty laboratory results i | neet the following effectia. |
|---|---|---|
| Liver | Chemistry Criteria Re | equiring Increased Follow-up |
| ALT or AST-absolute | ALT or AST $\geq 5 \times U$ | LN |
| ALT or AST Increase | ALT or AST $\geq 3 \times U$ | LN persists for ≥ 4 weeks |
| Bilirubin <sup>1,2</sup> | ALT or AST $\geq 3 \times U$ direct bilirubin) | LN <b>and</b> total bilirubin $\geq 2 \times \text{ULN}$ (> 35% |
| Cannot Monitor | ALT or AST $\geq 3 \times U$ .<br>4 weeks | LN and cannot be monitored weekly for |
| | | LN associated with symptoms (new or to be related to liver injury or hypersensitivity |
| Suggest | ed Actions, Monitorin | g, and Follow-up Assessments |
| Actio | ons | Follow-up Assessments |
| <ul> <li>Report the event to the Medical Monitor within 24 hours.</li> <li>Complete a Serious Adverse Event Report Form if the event also met the criteria for an SAE.<sup>2</sup></li> <li>Perform follow-up assessments as described in the Follow-up Assessment column.</li> <li>Monitor the participant until liver chemistry test abnormalities resolve, stabilize, or return to baseline.</li> <li>MONITORING:</li> <li>If ALT or AST ≥ 3 × ULN AND total bilirubin ≥ 2 × ULN:</li> </ul> | | <ul> <li>Viral hepatitis serology<sup>4</sup></li> <li>Obtain serum creatine phosphokinase (CPK), lactate dehydrogenase (LDH), gamma-glutamyltransferase [GGT], glutamate dehydrogenase [GLDH], and serum albumin.</li> <li>Fractionate bilirubin, if total bilirubin ≥ 2 × ULN.</li> <li>Obtain complete blood count with differential to assess eosinophilia.</li> <li>Record the appearance or worsening of clinical symptoms of liver injury, or hypersensitivity.</li> <li>Record use of concomitant medications (including acetaminophen, herbal</li> </ul> |
| <ul> <li>Repeat liver chemistry tests (include ALT,<br/>AST, ALP, and total bilirubin) and<br/>perform liver event follow-up assessments<br/>within 24 hours.</li> </ul> | | remedies, and other over-the-counter medications) on the concomitant medications eCRF. • Record alcohol use |

- Monitor participant twice weekly until liver chemistry test abnormalities resolve, stabilize, or return to baseline.
- A hepatology consultation is recommended.

## <u>If ALT or AST</u> $\ge$ 3 x <u>ULN AND total</u> <u>bilirubin < 2 x ULN:</u>

- Repeat liver chemistry tests (include ALT, AST, alkaline phosphatase, and total bilirubin) and perform liver chemistry follow-up assessments within 24 to 72 hours.
- Monitor participants weekly until liver chemistry abnormalities resolve, stabilize, or return to baseline.

If ALT or AST  $\geq$  3 x ULN AND total bilirubin  $\geq$  2 x ULN obtain the following in addition to the assessments listed above:

- Antinuclear antibody, antismooth muscle antibody, Type 1 antiliver kidney microsomal antibodies, and quantitative total immunoglobulin G (IgG), or gamma globulins
- Liver imaging (ultrasound, magnetic resonance, or computerized tomography) to evaluate liver disease
- Liver biopsy may be considered and discussed with local specialist if available, for instance:
  - In participants when serology raises the possibility of autoimmune hepatitis (AIH)
  - In participants when suspected druginduced liver injury (DILI) progresses or fails to resolve on withdrawal of study intervention
  - In participants with acute or chronic atypical presentation
- Report all assessments conducted to the Medical Monitor as they become available
- Serum bilirubin fractionation should be performed if testing is available. If serum bilirubin fractionation testing is unavailable, record the absence/presence of detectable urinary bilirubin on dipstick which is indicative of direct bilirubin elevations suggesting liver injury.
- 2. All events of ALT or AST >3 × ULN and total bilirubin > 2 × ULN (>35% direct bilirubin) may indicate severe liver injury (possible 'Hy's Law') and must be reported to sponsor in an expedited manner and as an SAE if SAE criteria met (excluding studies of hepatic impairment or cirrhosis).
- 3. New or worsening symptoms believed to be related to liver injury (such as fatigue, nausea, vomiting, right upper quadrant pain or tenderness, or jaundice) or hypersensitivity (such as fever, rash, or eosinophilia).
- 4. Includes: Hepatitis A immunoglobulin M (IgM) antibody; HBsAg and HBcAb; hepatitis C RNA; cytomegalovirus IgM antibody; Epstein-Barr viral capsid antigen IgM antibody (or if unavailable, heterophile antibody or monospot testing); and hepatitis E IgM antibody.

## 10.6. Appendix 6: Abbreviations

| Abbreviation | Definition |
|---|---|
| AE | Adverse Event |
| ADL | Activities of Daily Living |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Transaminase |
| AST | Aspartate Transaminase |
| ATC | Anatomical Therapeutic Chemical |
| b.i.d. | Twice Daily |
| BUN | Blood Urea Nitrogen |
| CFR | Code of Federal Regulations |
| CNS | Central Nervous System |
| CONSORT | Consolidated Standards of Reporting Trials |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders, 5 <sup>th</sup> Edition |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| eGFR | Estimated Glomerular Filtration Rate |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |
| FSH | Follicle-Stimulating Hormone |
| GAD | Generalized Anxiety Disorder |
| GCP | Good Clinical Practice |
| GLP | Good Laboratory Practice |

| HAM-D | Hamilton Depression Rating Scale |
|---|---|
| HBsAg | Hepatitis B Surface Antigen |
| hCG | Human Chorionic Gonadotropin |
| HCV | Hepatitis C Virus |
| HIV | Human Immunodeficiency Virus |
| HRT | Hormone Replacement Therapy |
| ICH | International Conference on Harmonization |
| ICF | Informed Consent Form |
| IMP | Investigational Medicinal Product |
| IND | Investigational New Drug |
| INR | International Normalized Ratio |
| IRB | Institutional Review Board |
| ITT | Intent-To-treat |
| IWRS | Interactive Web Response System |
| LSAS | Liebowitz Social Anxiety Scale |
| MCH | Mean Corpuscular Hemoglobin |
| MCV | Mean Corpuscular Volume |
| NCT | National Clinical Trial |
| PP | Per-Protocol |
| PTSD | Post-Traumatic Stress Disorder |
| QTcF | Fridericia-corrected QT Interval |
| QTL | Quality Tolerance Limit |
| RBC | Red Blood Cell |
| SAD | Social Anxiety Disorder |
| SAE | Serious Adverse Event |
| SAF | Safety (Population) |
| SAP | Statistical Analysis Plan |
| SCID-5-CT | Structured Clinical Interview for DSM-5 Disorders - Clinical Trials version |

| SD | Standard Deviation |
|---|---|
| SNRI | Serotonin Noradrenaline Reuptake Inhibitor |
| SoA | Schedule of Activities |
| SSPS-N | Self-Statements During Public Speaking (Negative Self-Statements subscale) |
| SSPS-State | Self-Statements During Public Speaking – State Version |
| SSPS-Trait | Self-Statements During Public Speaking – Trait Version |
| SSRI | Selective Serotonin Reuptake Inhibitor |
| STAI-State | Spielberger State-Trait Anxiety Inventory – State component |
| SUDS | Subjective Units of Distress Scale |
| TEAE | Treatment-Emergent Adverse Event |
| ULN | Upper Limit of Normal |
| US | United States |
| WBC | White Blood Cell |
| WHO-DD | World Health Organization Drug Dictionary |
| WOCBP | Woman of Childbearing Potential |
| WONCBP | Woman of Non-childbearing Potential |

| 4 | 4 | T) ( |
|---|----|----------------|
| • | 1. | . References |
| 1 | | . IXCICI CHCCS |



FDA Drug Safety Communication 23<sup>rd</sup> Sep 2020: <a href="https://www.fda.gov/media/142368/download">https://www.fda.gov/media/142368/download</a>

Graeff FG, Parente A, Del-Ben CM, Guimarães FS. Pharmacology of human experimental anxiety. Braz J Med Biol Res. 2003 Apr;36(4):421-32.

Heimberg RG. Cognitive-behavioral therapy for social anxiety disorder: current status and future directions. Biol Psychiatry. 2002 Jan 1;51(1):101-8.

Heimberg RG, Liebowitz MR, Hope DA, Schneier FR, Holt CS, Welkowitz LA, et al. Cognitive behavioral group therapy vs phenelzine therapy for social phobia: 12-week outcome. Arch Gen Psychiatry. 1998 Dec;55(12):1133-41.

Hofmann SG, Dibartolo PM. An instrument to assess self-statements during public speaking: scale development and preliminary psychometric properties. Behav Ther. 2000;31(3):499-515.



Osório FL, Crippa JA, Loureiro SR. Validation of the state version of the Self-Statement during Public Speaking Scale. Braz J Psychiatry. 2013 Mar;35(1):63-6. doi: 10.1016/j.rbp.2012.02.009. PMID: 23567602



Wolpe J. The practice of behavior therapy. New York: Pergamon Press; 1969.